CLINICAL TRIAL: NCT03324646
Title: Evaluation of a Novel PET Radioligand to Image Cyclooxygenase-1 (COX-1)
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170179; 17-M-0179
Record Dates: First submitted 2017-10-27; First posted 2017-10-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Normal Physiology
Keywords: Research; Brain; Inflammation; Natural History
MeSH Terms: conditions — Inflammation | interventions — 11C-PS13

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- controls: healthy subjects
  Interventions: Drug: [11C]PS13

INTERVENTIONS:
Drug: [11C]PS13 — A novel PET ligand to selectively image COX-1

SUMMARY:
Background:

A radioligand is a radioactive substance that is used to diagnose diseases. A new ligand is called [11C]PS13. This has a small amount of radioactivity that can be detected by a positron emission tomography (PET) scan. If this ligand works well in this study, researchers may be able to use it to better understand and diagnose brain disorders.

Objectives:

To evaluate if [11C]PS13 can measure its receptor, which is involved in inflammation. To see if researchers get the same results when scanning a person twice.

Eligibility:

Healthy people ages 18 and older who are in Protocol 01-M-0254.

Design:

This study requires three visits of 2-5 hours each.

Participants will have 2 PET scans with [11C]PS13.

A needle will guide a small plastic tube (catheter) into an arm vein. The needle will be removed, leaving only the catheter in the vein. The ligand will be injected through the catheter.

The PET scanner is shaped like a doughnut. Participants will lie on a bed that slides in and out of the scanner.

Participants will wear a molded a plastic mask that fits the head.

Another catheter will be put into an artery at the wrist or elbow area.

Vital signs will be monitored during the PET scan. Participants will have a test during the PET scan to monitor heart function.

Participants will have blood and urine tests.

Participants will have 1 magnetic resonance imaging (MRI) scan. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder.

DETAILED DESCRIPTION:
Objective

The cyclooxygenase (COX) system is implicated in the pathophysiology of brain diseases, including Alzheimer s disease and depression, and is a potential biomarker for neuroinflammation. COX is the rate-limiting enzyme in the synthesis of prostaglandins from arachidonic acid and exists as two primary isoforms COX-1 and COX-2. Our laboratory recently developed [(11)C]PS13, a novel PET ligand to selectively image COX-1, and initial PET scans in monkey demonstrated that [11C]PS13 is a promising ligand.

This study has two primary objectives. First, we will determine whether the uptake of [(11)C]PS13 in brain and periphery reflects the distribution of COX-1, as demonstrated by blocking with a COX-1 preferential drug (aspirin or ketoprofen) and/or no effect with a COX-2 selective drug (celecoxib). Second, we will measure the test/retest reproducibility of brain uptake quantified by compartmental modeling and using arterial and/or venous blood samples.

Study Population

Healthy adult volunteers (aged 18 years or older) will have either whole body imaging (n = 41) or brain imaging (n = 20).

Design

Phase 1: We will begin with whole body scanning in a single human subject using up to 10 mCi. The aim of this first scan will be to detect a tracer that disproportionately accumulates in a single radiosensitive organ, such as the gonads. If we confirm that radioactivity is fairly widely distributed in the body, higher activities may be injected.

Phase 2:Thirty healthy subjects will have three whole body imaging PET scans using 20 mCi of [11C]PS13. Scan 1 will serve as the baseline scan for comparison to enzyme occupancy studies and will provide dosimetry information. Scan 2 will be an enzyme occupancy study using the COX-2 selective antagonist celecoxib. Scan 3 will be an enzyme occupancy study using the COX-1 preferential antagonist aspirin. Ten healthy subjects will have two whole body imaging PET scans using 20 mCi of [11C]PS13. Scan

1 will serve as the baseline scan, and scan 2 will be an enzyme occupancy study using another potent COX-1 antagonist ketoprofen.

Phase 3: We will perform 15 test retest kinetic brain imaging PET studies with arterial and/or venous blood sampling and 5 test retest brain PET studies with both arterial and venous blood sampling, using a 20 mCi dose of [(11)C]PS13.

Outcome Measures

For whole body imaging, organ uptake will be quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight. Blockade by aspirin, ketoprofen, and celecoxib will be expressed as a percentage of the baseline scan in each subject and plotted relative to the plasma concentration of the drug at time of the PET scan. For dedicated brain imaging, uptake will be quantified as distribution volume (VT) calculated with compartmental modeling and serial concentrations of parent radioligand in arterial and/or

venous plasma.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 years or older.
* Able to provide informed consent.
* Medically and psychiatrically healthy.
* Enrolled in 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17-M-0181, Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies".

EXCLUSION CRITERIA All phases

* Because non-steroidal anti-inflammatory drugs (NSAIDs) inhibit COX-1 and/or COX-2, subjects should not have taken NSAIDs for two weeks prior to the PET scan. In addition, aspirin must not have been taken in the prior month, as aspirin irreversibly inhibits COX.
* Clinically significant laboratory abnormalities based on tests performed under screening protocol 01-M-0254 or 17-M-0181 and specified in Section 4.c Screening.
* Any current Axis I diagnosis, based on interview and self-reporting performed under screening protocol 01-M-0254 or 17-M-0181.
* HIV infection.
* History of medical or neurologic illness or injury with the potential to affect study data interpretation.
* Recent exposure to radiation related to research (i.e. PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breastfeeding.
* Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not

exclusion criteria, unless that use impairs function of daily life..

* Current use of psychiatric medications.
* NIMH employees and staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

EXCLUSION CRITERIA Phase 2:

* Because aspirin and celecoxib require an acidic environment to be absorbed in the stomach, we will exclude those who have taken proton pump inhibitor (PPI) drugs, H-2 receptor antagonist drugs, and antacid drugs in the last two weeks.
* additional contraindications to taking COX-1 or COX-2 inhibitors include:

  * history of hypersensitivity reaction to COX inhibitors history of aspirin- or NSAID-induced asthma.
  * history of upper or lower gastrointestinal bleeding, gastritis, peptic ulcer disease, or gastroesophageal reflux disease (GERD).
  * coagulation disorder.
  * thrombocytopenia.
  * G6PD deficiency.
  * history of gout.
  * history of hepatic or renal impairment.
  * history of cardiovascular disease or presence of cardiovascular risk factors such as hypertension.

EXCLUSION CRITERIA Phase 3:

* Artery check for art line
* Unable to have an MRI scan

NIH employees are eligible to participate. NIMH employee participation is guided by intramural institute policy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
PET tracer update | during PET scan
  For whole body imaging, organ uptake will be quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight. Blockade by aspirin, ketoprofen, and celecoxib will be expressed as a percentage of the baseline scan in each subject and plotted relative to the plasma concentration of the drug at time of the PET scan. For dedicated brain imaging, uptake will be quantified as distribution volume (VT) calculated with compartmental modeling and serial concentrations of parent radioligand in arterial and/or venous plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kim MJ, Lee JH, Juarez Anaya F, Hong J, Miller W, Telu S, Singh P, Cortes MY, Henry K, Tye GL, Frankland MP, Montero Santamaria JA, Liow JS, Zoghbi SS, Fujita M, Pike VW, Innis RB. First-in-human evaluation of [11C]PS13, a novel PET radioligand, to quantify cyclooxygenase-1 in the brain. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3143-3151. doi: 10.1007/s00259-020-04855-2. Epub 2020 May 12. PMID 32399622
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-M-0179.html